CLINICAL TRIAL: NCT06829199
Title: A Phase 2, Umbrella Study to Evaluate the Safety, Tolerability, and Clinical Activity of Investigational Agents for Newly Diagnosed, High-Risk, Early-Stage Triple-Negative Breast Cancer
Brief Title: A Clinical Study of Boserolimab (MK-5890) With Pembrolizumab and Chemotherapy in People With Early Triple-Negative Breast Cancer (MK-5890-003)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Since patients were not recruited yet, we would mark this as a Withdrawn status per the NIH definition of that status. Study halted prematurely, prior to enrollment of first participant.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5890-003; MK-5890-003 (Other: MSD); 2024-517505-87-00 (Registry Identifier: EU CT); U1111-1312-3982 (Registry Identifier: UTN)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Early Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Breast cancer; Neoadjuvant; Boserolimab; Pembrolizumab; Umbrella study
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Paclitaxel; Carboplatin; Doxorubicin; Epirubicin; Cyclophosphamide; Capecitabine; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+ Paclitaxel+ Carboplatin (Active Comparator): Participants will receive pembrolizumab PLUS paclitaxel PLUS carboplatin followed by pembrolizumab PLUS doxorubicin hydrochloride or epirubicin hydrochloride and cyclophosphamide as neoadjuvant therapy prior to surgery. In adjuvant therapy participants will receive pembrolizumab PLUS optional additional adjuvant treatment of physician's choice (TPC), capecitabine or olaparib.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin (hydrochloride); Drug: Epirubicin Hydrochloride; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib (if approved/available locally)
- Pembrolizumab+Boserolimab+Paclitaxel+ Carboplatin (Experimental): Participants will receive pembrolizumab PLUS boserolimab PLUS paclitaxel PLUS carboplatin followed by pembrolizumab PLUS doxorubicin hydrochloride or epirubicin hydrochloride and cyclophosphamide PLUS boserolimab as neoadjuvant therapy prior to surgery. In adjuvant therapy participants will receive pembrolizumab PLUS optional additional adjuvant treatment of physician's choice (TPC), capecitabine or olaparib.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin (hydrochloride); Biological: Boserolimab; Drug: Epirubicin Hydrochloride; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib (if approved/available locally)

INTERVENTIONS:
Biological: Pembrolizumab — Neoadjuvant therapy - 200 mg intravenous (IV) infusion every 3 weeks (Q3W) for up to approximately 24 weeks Adjuvant therapy - 200 mg IV infusion Q3W or 400 mg IV infusion every 6 weeks (Q6W) for up to approximately 30 weeks.
  Other Names: MK-3475; Keytruda®; SCH 900475
Drug: Paclitaxel — 80 mg/m^2 by IV infusion every week for up to 12 weeks.
Drug: Carboplatin — AUC 1.5 mg/mL/min by IV infusion every week for up to 12 weeks.
Drug: Doxorubicin (hydrochloride) — 60 mg/m^2 by IV infusion Q3W for up to 12 weeks.
Biological: Boserolimab — 30 mg by IV infusion every 6 weeks (Q6W) for up to 12 Weeks.
  Other Names: MK-5890
  Arms: Pembrolizumab+Boserolimab+Paclitaxel+ Carboplatin
Drug: Epirubicin Hydrochloride — 90 mg/m^2 by IV infusion every 3 weeks (Q3W) for up to 12 weeks.
Drug: Cyclophosphamide — 600 mg/m^2 by IV infusion every 3 weeks (Q3W) for up to 12 weeks.
Drug: Capecitabine — 1000 mg/m^2 to 1250 mg/m^2 by oral administration twice a day (2 weeks on and 1 week off) for up to approximately 24 weeks.
Drug: Olaparib (if approved/available locally) — 300 mg by oral administration twice a day for up to approximately 52 weeks.

SUMMARY:
Researchers want to learn if giving boserolimab (MK-5890) with standard treatment (pembrolizumab and chemotherapy) before surgery can help treat triple negative breast cancer (TNBC). The goals of this study are to learn about the safety of boserolimab given with standard treatment before surgery and to learn if people tolerate it and how many people have no signs of cancer in the tissues and lymph nodes removed during surgery.

DETAILED DESCRIPTION:
The umbrella design of this study provides the framework to evaluate the safety, tolerability and clinical activity of different investigational agents in participants with newly diagnosed, high-risk, early-stage TNBC who might benefit from adding these investigational agents to pembrolizumab plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has previously untreated high-risk, early-stage, non-metastatic (M0) breast cancer (BC), defined as tumor stage T1c, nodal stage N1-2, or tumor stage T2-4, nodal stage N0-2
* Has provided a core needle biopsy for tissue diagnosis of the current breast cancer less than 29 days prior to the date of informed consent
* Has centrally confirmed diagnosis of BC that is triple-negative based on the American Society of Clinical Oncology/College of American Pathologists guidelines
* Has Eastern Cooperative Oncology Group performance status of 0 or 1 performed within 28 days before treatment randomization
* Has left ventricle ejection fraction of ≥50% as assessed by echocardiogram or multigated acquisition scan performed at screening
* Has a history of exposure to anthracycline; participants can be eligible after completion of a Sponsor consultation form, if cumulative lifetime doses are as follows: Doxorubicin <100 mg/m2, Epirubicin <180 mg/m2, Mitoxantrone <40 mg/m2, Idarubicin <22.5 mg/m2. Note: If another anthracycline or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of 100 mg/m2 of doxorubicin

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has documented Grade ≥2 peripheral neuropathy
* Has uncontrolled or significant cardiovascular disease
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein-4 [CTLA-4], OX-40 [cluster of differentiation (CD) 134], or CD137)
* Has received any prior treatment, including radiation, systemic therapy, and/or definitive surgery for currently diagnosed breast cancer
* Has received prior systemic anticancer therapy
* Has undergone excisional biopsy of the primary tumor and/or axillary lymph node dissection prior to study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has active autoimmune disease that has required systemic treatment in the past 2 years with need for disease modifying agents such as corticosteroids or immunosuppressive drugs
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has severe hypersensitivity (Grade ≥3) to pembrolizumab, any investigational agent or study intervention, any of its excipients, and/or to another biologic therapy
* Has a history of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-26 (Estimated); Primary Completion 2029-01-18 (Estimated); Study Completion 2031-03-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with one or more adverse events (AEs) | Up to approximately 34 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Number of participants who discontinue study intervention due to an AE | Up to approximately 27 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Pathological complete response (pCR) rate at the time of definitive surgery | Up to approximately 9 months
  pCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy per current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
pCR-no ductal carcinoma in situ (DCIS) rate at the time of definitive surgery | Up to approximately 9 months
  pCR-no ductal carcinoma in situ (DCIS) (ypT0 ypN0) is defined as the absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy per current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery.
Event-Free Survival (EFS) | Up to approximately 72 months
  EFS is defined as the time from randomization to disease progression that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 72 months
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Optum Care Cancer Center ( Site 0004), Las Vegas, Nevada, United States
- National Cheng Kung University Hospital ( Site 0901), Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/